CLINICAL TRIAL: NCT06489769
Title: Prevalence of Opioid Misuse in Patients with Cancer
Brief Title: Opioid Misuse in Patients with Cancer
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Geana P Kurita, Professor, Rigshospitalet, Denmark
Other Study IDs: 100845
Record Dates: First submitted 2024-06-27; First posted 2024-07-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Opioid Use; Opioid Misuse; Pain; Cancer Pain
MeSH Terms: conditions — Neoplasms; Opioid-Related Disorders; Pain; Cancer Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The success of opioid treatment in terminally ill cancer patients set the stage for extending the same treatment principles to the treatment of all chronic pain conditions including chronic non-cancer pain and chronic pain in cancer, where survival and long-standing chronic disease trajectories are getting more prevalent due to increasing survival rates. In this context, opioid misuse as such has been highly neglected - especially in palliative care, but also in cancer pain management in general. Previous studies have explored the literature on opioid misuse among adult cancer patients, noting that the available evidence is still in its early stages. Limited prospective studies with a wide range of definitions and methodologies for assessing misuse exist. Therefore, it seems highly relevant and justified to study the prevalence of opioid misuse risk in patients with cancer. The hypothesis of this study is that opioid misuse is not uncommon in Danish patients in treatment with opioids for cancer-related pain. Thus, the prevalence of opioid misuse risk among patients with cancer in Danish palliative care units will be investigate.

DETAILED DESCRIPTION:
This is a prospective and cross-sectional study, in which opioid misuse is defined according to National Institute on Drug Abuse (USA) as the use of prescription opioids in a manner other than as directed by a doctor (e.g., for other purpose than pain relief, in greater amounts, more frequently, longer, using someone else's prescription). The aims are:

1. Investigate the prevalence of opioid misuse risk by the Pain Medication Questionnaire (PMQ) and the Opioid Risk Tool (ORT) among patients with cancer in palliative care units in Denmark.
2. Determine whether there is a correlation between the PMQ and ORT scores and opioid consumption, use of short-acting opioids (prn-dosing), tobacco smoking, alcohol consumption, previous consumption of illicit drugs and/or consumption of benzodiazepines and benzodiazepine-like hypnotics, and information provided by the physician regarding the patient's opioid misuse.
3. Investigate the association between opioid misuse risk (PMQ and ORT scores), depression and anxiety (Patient Health Questionnaire for Depression and Anxiety, PHQ-4), and health-related quality of life (EORTC-QLQ-C15-PAL).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥ 18 years,
* patients who are treated with opioids due to cancer-related pain.

Exclusion Criteria:

* Patients who do not master the Danish language in speech and writing,
* Patients who have severe cognitive dysfunction,
* Patients who are not treated with opioids,
* Patients who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Section of Palliative Medicine at Rigshospitalet.
  Patients can participate if ≥ 18 years and able to communicate in Danish.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Medication Questionnaire (PMQ) | Baseline
  PMQ consists of 26 questions assesses the risk of opioid abuse in people with non-oncological chronic pain. The answers are given on a 5-point Likert scale. Total score varies between 0 and 104 points.
Opioid Risk Tool (ORT) | Baseline
  ORT consists of a 5-question screening instrument assessing the risk for opioid abuse among individuals prescribed opioids for treatment of chronic pain.

SECONDARY OUTCOMES:
Pain diagnosis | Baseline
  Categories: nociceptive somatic, nociceptive visceral, neuropathic, nociplastic, nociceptive +somatic (mixed).
Pain duration | Baseline
  In months.
Pain localization | Baseline
  Categories: head/face/mouth/neck, up limbs, lower limbs, thorax, abdomen, low back/gluteus/coccyx/pelvis.
Pain intensity | Baseline
  Numerical scale from 0 (no pain) to 10 (worst pain).
Opioids | Baseline
  Patient consumption of opioids. Name, dose and duration of treatment will be recorded. When treated with opioids, doses are converted to oral morphine equivalents. Data will be collected from patients electronic records.
Benzodiazepines | Baseline
  Patient consumption of benzodiazepines: Name, dose and duration of treatment will be recorded. Data will be collected from patients electronic records.
Hypnotics | Baseline
  Patient consumption of Hypnotics: Name, dose and duration of treatment will be recorded. Data will be collected from patients electronic records.
Alcohol | Baseline
  Alcohol consumption (number of drinks per week). The following question will be used to assess the amount of alcohol intake: ''How many alcoholic drink glasses did you have each day last week? We'll start with yesterday and take one day at a time''.
Tobacco | Baseline
  Tobacco use (number of cigarettes, cigars and/or pipe tobacco per day). Smoking behaviour will be assessed by asking the respondent whether they smoked or not, and smokers were asked about their average daily number of smoked cigarettes. Heavy smokers were defined as individuals smoking at least 15 cigarettes a day
Patient Health Questionnaire-4 (PHQ-4) | Baseline
  The validated two-item ultra-brief screeners for depression (PHQ-2) and anxiety (GAD-2) were combined to constitute the PHQ-4. PHQ-4 is a reliable and valid instrument for screening depressive and anxiety symptoms, both for the clinical and nonclinical populations. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 - Palliative Care (EORTC-QLQ-C15-PAL) | Baseline
  The EORTC-QLQ-C15-PAL is a 'core questionnaire' for use in palliative care and focuses on frequent symptoms, emotional and physical function, and global health status/ quality of life. It includes 15 items with two multi- item functional scales (physical and emotional functioning), two multi-item symptom scales (fatigue and pain) and a five single item symptom scale (dyspnoea, appetite loss, nausea and vomiting, insomnia, and constipation). One item addresses the global health status/ quality of life. The responses are on a 1-4-point Likert scale for all items ranging from 1 (not at all) to 4 (very much), except for one item measuring global health status/quality of life ranging from 1 (very poor) to 7 (excellent). For functioning scales, 100 represents good functioning with no problems. For symptom scales, 100 represents a high degree of symptom burden.
The patients' self-assessed health | Baseline
  To assess the patients' self-assessed health the following question will be used: 'How is your health overall? ´ The respondents rate excellent, very good, good, less good or poor. The question has been used in previous large national surveys of the general population in Denmark.
Information provided by the physician regarding the patient's opioid misuse | 1 month after baseline
  The physician treating the patient at the palliative care unit will be asked regarding the patient's potential opioid misuse. The physician will receive written information outlining the operational definition of opioid misuse applied in this study, followed by a closed question: 'In your clinical evaluation, is the patient (identification information: name) an opioid misuser?' The response options are 'Yes,' 'No,' 'Maybe,' and 'I do not know.'

OTHER OUTCOMES:
Sex | Baseline
  Categories male, female.
Age | Baseline
  Complete years in number.
Marital status | Baseline
  Categories; single (unmarried), married, cohabitating, separated/divorced, widow/widower.
Education status | Baseline
  Categories, basic school, upper secondary or vocational school, higher education.
Schooling | Baseline
  Number of years of formal education.
Income | Baseline
  Categories in Danish Krone (DKK): <200.000 DKK, 200.000-500.000 DKK, >500.000 DKK
Occupational status | Baseline
  Categories: working/studying, retired, on sick leave.

CONTACTS AND LOCATIONS:
Overall Officials: Geana Kurita, PHD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, København Ø., Denmark

IPD SHARING:
Plan to Share IPD: No